CLINICAL TRIAL: NCT05964036
Title: Personalized Brain Functional Sectors (pBFS)-Guided DMPFC With High-dose rTMS for Treatment-resistant Depressive Disorder: a Randomized, Double-blind, Sham-controlled Trial
Brief Title: pBFS-guided High-dose TMS Over DMPFC for Treatment-resistant Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changping Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPLMDDHidoseDM
Record Dates: First submitted 2023-07-12; First posted 2023-07-27 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-07

CONDITIONS: Depression; Major Depressive Disorder; Severe Depression
Keywords: transcranial magnetic stimulation, rTMS; DMPFC; pBFS; precision target
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active TMS (Experimental): active iTBS coupled with medical therapy
  Interventions: Device: active TMS
- sham TMS (Sham Comparator): Sham iTBS coupled with medical therapy
  Interventions: Device: sham TMS

INTERVENTIONS:
Device: active TMS — Participants will receive 10 sessions per day of 1800 pulses per session, lasting for 5 days. Individualized target in the DMPFC will be generated using the pBFS method
  Arms: active TMS
Device: sham TMS — The parameters in the sham arm are the same as in the active stimulation group. Stimulation was delivered by the same device as the active group fitted with a sham coil
  Arms: sham TMS

SUMMARY:
The investigators aim to evaluate the safety and efficacy of pBFS-guided DMPFC target and high-dose rTMS therapy for the treatment of patients with treatment-resistant depression

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established therapy for treatment-resistant depression. Currently, the FDA cleared the SAINT Neuromodulation System for the treatment of Treatment-Resistant Depression(TRD) over the left dorsolateral prefrontal cortex (DLPFC). This methodology has been effective in a short period of time for treatment-resistant depression. However, some patients may not be able to persist in completing the treatment because they cannot bear the pain during treatment. The dorsomedial prefrontal cortex (DMPFC) region is relatively posterior, and DMPFC as an intervention target has been proven to have antidepressant effects, and patients have better pain tolerance during treatment, which can be used as an alternative to DLPFC target, so it is urgent to explore the effectiveness and safety of high-dose iTBS targeting DMPFC in the treatment of depression.

After being informed about the study and potential risks. All patients giving written informed consent will undergo a screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a blind manner in a 2:1 ratio to the active-rTMS group, and sham-rTMS group. Then all participants will undergo a 5-day rTMS modulation followed by two-week and four-week follow-up visits. Participants will keep a stable treatment regime during treatment and the four-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of depressive disorder, recurrent episodes;
* A total score of at least 20 on the HAMD-17 and Montgomery-Asberg Depression Rating Scale;
* Aged 18-65 years, female or male;
* Inadequate response to at least one antidepressant trial of adequate doses and duration;
* The MSM (Maudsley Staging Method) score ≥ 7;
* Stable antidepressant regimen for at least 4 weeks before treatment;
* Understand the trial and sign the informed consent.

Exclusion Criteria:

* Meet DSM-5 diagnostic criteria for other mental disorders (such as schizophrenia spectrum disorders, bipolar and related disorders, neurodevelopmental disorders, neurocognitive disorders, or depressive disorders due to substances and/or medications, depressive disorders due to other medical problems, etc.);
* Patients with a cardiac pacemaker, cochlear implant, or other metal foreign body and any electronic equipment implanted in the body, patients with claustrophobia and other contraindications to magnetic resonance scanning, and patients with contraindications to rTMS treatment;
* Patients with serious or unstable diseases of the cardiovascular, liver, kidney, blood, endocrine, neurological system, and other systems or organs, especially those with organic brain diseases (such as ischemic stroke, cerebral hemorrhage, brain tumor, etc.) and a history of severe brain trauma as judged by the researcher;
* History of epilepsy (presence of at least 2 uninduced seizures more than 24 hours apart, or diagnosis of the epileptic syndrome, or seizures within the past 12 months); Or currently received medications or other treatments that will lower the seizure threshold;
* History of ECT, rTMS, VNS, DBS, tDCS, light therapy, or other physical therapy related to mental illness within 3 months;
* Currently receiving or planning to start formal cognitive or behavioral therapy, or systemic psychological therapy (interpersonal therapy, dynamic therapy, cognitive behavioral therapy, etc.) during the trial.
* Substance abuse or dependence (including alcohol, drugs, and other psychoactive substances) in the past 1 year;
* The female of childbearing potential who plans to become pregnant during the trial, and that is pregnant or breastfeeding.
* Patients in any clinical trials of other drugs or physical therapy within 1 month before the screening.
* First-degree relatives have bipolar affective disorder.
* Difficulty or inability to engage in normal communication, understand or follow instructions, and cooperate with treatment and evaluators.
* Investigators think that was inappropriate to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
change in Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline, Day 5
  The MADRS is a validated instrument stratifying the severity of depressive episodes in adults. The MADRS has an overall score ranging from 0 (no depression) to 60 (worst depression).

SECONDARY OUTCOMES:
Change in MADRS | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment
  A provider-administered questionnaire was used to assess remission and recovery from depression. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The MADRS has an overall score range from 0-60, with higher scores corresponding to higher levels of depression
Change in Hamilton Depression Scale (HAMD-17) | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment
  A provider-administered questionnaire was used to assess remission and recovery from depression. The Hamilton Depression Rating Scale (HAMD) is the most widely used clinician-administered depression assessment scale. The Ham-17 version consists of 17 items assessing mood, guilt, general somatic symptoms, work and activities, anxiety, and slowness of thought and speech. Each item is scored on a scale of 0 to 4, except for the somatic, sleep, and insight items which are scored 0 to 2. On the HAMD-17 there can be a total score of 52. Higher scores represent higher depression severity.
Change in Quick Inventory of Depressive Symptomatology Self-Report (QIDS_SR) | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment
  A provider-administered questionnaire was used to assess remission and recovery from depression. The 16-item QIDS_SR is a widely used self-report instrument covering depressive symptoms incorporating nine Diagnostic and Statistical Manual of Mental Disorder-IV (DSM-IV) diagnostic criteria for major depressive disorders. Each item is scored on a scale of 0 to 4. Higher scores represent higher depression severity.
cognitive change in Digit Symbol Substitution Test (DSST) | Baseline, Day 5 (Immediate Post-treatment)
  Cognitive scores are measured using Chinese brief cognitive test (C-BCT), the DSST equires a subject to match symbols to numbers according to a key located on the top of the page
cognitive change in continuous performance test (CPT) | Baseline, Day 5 (Immediate Post-treatment)
  CPT from the C-BCT measures a person's sustained and selective attention
cognitive change in Trail-Making Test (TMT) | Baseline, Day 5 (Immediate Post-treatment)
  The TMT test from the C-BCT can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning
cognitive change in Digit Span Test (DST) | Baseline, Day 5 (Immediate Post-treatment)
  DST from the C-BCT is a measure of verbal short term and working memory that can be used in two formats, Forward Digit Span and Reverse Digit Span
Safety estimated using SSI | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment
  Scale for Suicide Ideation (SSI) measures suicide ideation
Safety estimated using YMRS | Baseline, Day 5 (Immediate Post-treatment), 14 days Post-treatment, 28 days Post-treatment
  Young Mania Rating Scale(YMARS) measures mania

CONTACTS AND LOCATIONS:
Overall Officials: hesheng Liu, Study Chair — Changping Laboratory
Locations (1):
- Hebei Mental Health Center, Baoding, Hebei, China